CLINICAL TRIAL: NCT06846840
Title: Effect of Ketone Esters Ingested During Recovery on Metabolism and Subsequent Exercise Capacity
Brief Title: Ketone Esters and Metabolism During Recovery from Endurance Exercise
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Professor of Nutrition and Metabolism, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 5202-6834
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Exercise; Metabolism
MeSH Terms: conditions — Motor Activity | interventions — formic acid 4-(3-oxobutyl)phenyl ester

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLACEBO (Placebo Comparator): Energy matched placebo containing medium-chain triglycerides and bitter taste
  Interventions: Dietary Supplement: Placebo
- KETONE (Experimental): Beta-hydroxybutyrate monoester
  Interventions: Dietary Supplement: Ketone ester

INTERVENTIONS:
Dietary Supplement: Ketone ester — 0.29 g per kilogram body mass per hour of ketone monoester (R)-3-hydroxybutyrate (R)-3-hydroxybutyl
  Arms: KETONE
Dietary Supplement: Placebo — Medium chain triglycerides and bitter tastant (Bitrex)
  Arms: PLACEBO

SUMMARY:
Infusion of beta-hydroxybutyrate can suppress endogenous glucose production, which may result in increased net liver glycogen storage. If ketone esters exert similar effects, then the increase in liver glycogen storage may have implication for recovery from exercise and subsequent exercise performance.

The aim of this study is to assess the effects of ketone esters ingested during recovery from exercise, on metabolism and subsequent exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* VO2max ≥ 45mL.kg-1.min-1
* Weekly aerobic training > 3hours.
* 2years running experience.
* BMI < 30kg/m2

Exclusion Criteria:

* <18yrs or >60yrs of age
* Habitual smoker within last 5 years.
* History of uncontrollable metabolic or respiratory disease.
* Currently taking medication, following a low carbohydrate or ketogenic diet, or consuming nutritional ketone supplements.
* History of Irritable Bowel Syndrome

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Glucose concentrations | 240 minutes
  Blood glucose concentrations during the recovery period (240 minutes)

SECONDARY OUTCOMES:
Non-oxidative fate of ingested sucrose | 240 minutes
  Non-oxidative fate of ingested glucose measured by appearance of 13C on breath CO2 from high 13C sucrose ingested during recovery
Exercise capacity | 240 minutes
  Time to exhaustion running at 70% of maximal aerobic capacity after the recovery period

OTHER OUTCOMES:
Blood beta-hydroxybutyrate concentrations | 240 minutes
  Blood beta-hydroxybutyrate concentrations throughout the 240 minute recovery
Urinary urea | 240 minutes
  Urea in urine, determined by urea concentration multiplied by total urine output during the 240 minutes of recovery
Blood lactate concentrations | 240 minutes
  Blood lactate concentrations during 240 minutes of recovery
Plasma insulin concentrations | 240 minutes
  Plasma insulin concentrations during 240 minutes of recovery
Blood pH | 240 minutes
  Blood pH during 240 minutes of recovery
Blood bicarbonate | 240 minutes
  Blood bicarbonate concentrations during 240 minutes of recovery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Plan is to share individual deidentied data on a public repository such as Mendeleydata.